CLINICAL TRIAL: NCT01110798
Title: Colonic J-Pouch Reconstruction Versus Straight Colorectal Anastomosis After Low Anterior Resection for Rectal Cancer: Impact on Anastomotic Leak, Bowel Function and Quality of Life
Brief Title: J-Pouch Colorectal Anastomosis or Straight Colorectal Anastomosis in Treating Patients With Rectal Cancer Who Have Undergone Surgery to Remove the Tumor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera di Padova (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000671070; USP-1935P; EU-21032
Record Dates: First submitted 2010-04-23; First posted 2010-04-27 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2011-02

CONDITIONS: Colorectal Cancer; Gastrointestinal Complications; Perioperative/Postoperative Complications
Keywords: perioperative/postoperative complications; gastrointestinal complications; adenocarcinoma of the rectum; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Postoperative Complications; Rectal Neoplasms

INTERVENTIONS:
Other: intraoperative complication management/prevention
Procedure: assessment of therapy complications
Procedure: gastrointestinal complications management/prevention
Procedure: quality-of-life assessment
Procedure: therapeutic conventional surgery

SUMMARY:
RATIONALE: It is not yet known whether a J-pouch colorectal anastomosis is more effective than a straight colorectal anastomosis in treating patients with rectal cancer who have undergone surgery to remove the tumor.

PURPOSE: This randomized clinical trial is studying J-pouch colorectal anastomosis to see how well it works compared with straight colorectal anastomosis in treating patients with rectal cancer who have undergone surgery to remove the tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess whether the incidence of major anastomotic leak after low anterior resection, in patients with rectal cancer, is reduced by using the J-pouch reconstruction vs straight colorectal anastomosis.

Secondary

* To compare the global anastomotic leak (major and minor) rate, the incidence of other complications in addition to anastomotic leak, and the functional outcome and the quality of life in these patients.
* To describe, in the J-pouch reconstruction group, the feasibility of the colonic J-pouch.

OUTLINE: Ths is a multicenter study. Patients are stratified according to clinical center, gender (male vs female), and neoadjuvant treatment types. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo a total mesorectal excision with a low anterior rectal resection followed by a mechanical straight stapled colorectal anastomosis.
* Arm II: Patients undergo a total mesorectal excision with a low anterior rectal resection followed by a mechanical J-pouch stapled anastomosis reconstruction.

Quality of life is assessed periodically using EORTC Quality of Life Questionnaires (EORTC QLQ-C30 and -CR38), and the MSKCC Bowel Function Questionnaire.

After completion of study treatment, patients are followed at 1, 6, 12, and 24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed rectal adenocarcinoma meeting the following criteria:

  * Mid and/or low rectal cancer
  * Tumor site ≤ 11 cm from anal verge
  * Must have a temporary stoma (ileostomy or colostomy)
* Must be scheduled for a total mesorectal excision with a low anterior rectal resection and mechanic colorectal anastomosis that is potentially curative or with a microscopic residual resection (R0-R1)
* No locally recurrent disease
* No distant metastasis

PATIENT CHARACTERISTICS:

* Must be able to understand the study

PRIOR CONCURRENT THERAPY:

* No prior handsewn coloanal anastomosis
* No prior colonic resection
* No prior surgery for local recurrence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Major anastomotic leak rate

SECONDARY OUTCOMES:
Percentage of the colonic J-pouch reconstruction performed with respect to the total number of patients selected for the J-pouch treatment arm
Global anastomotic leak rate
Anastomotic complications rate in addition to anastomotic leak
Bowel function, fecal incontinence, and quality of life, evaluated with validated questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Donato Nitti, MD, Principal Investigator — Azienda Ospedaliera di Padova
Locations (4):
- Italy (4):
  - Universita Degli Studi di Florence - Policlinico di Careggi, Florence
  - Fondazione Istituto Nazionale dei Tumori, Milan
  - Azienda Ospedaliera di Padova, Padua
  - Ospedale Civile Di San Vito Al Tagliamento, San Vito Al Talgliamento

REFERENCES:
- [Derived] Gavaruzzi T, Pace U, Giandomenico F, Pucciarelli S, Bianco F, Selvaggi F, Restivo A, Asteria CR, Morpurgo E, Cuicchi D, Jovine E, Coletta D, La Torre G, Amato A, Chiappa A, Marchegiani F, Rega D, De Franciscis S, Pellino G, Zorcolo L, Lotto L, Boccia L, Spolverato G, De Salvo GL, Delrio P, Del Bianco P. Colonic J-Pouch or Straight Colorectal Reconstruction After Low Anterior Resection For Rectal Cancer: Impact on Quality of Life and Bowel Function: A Multicenter Prospective Randomized Study. Dis Colon Rectum. 2020 Nov;63(11):1511-1523. doi: 10.1097/DCR.0000000000001745. PMID 33044292
- [Derived] Jakob MO, Haltmeier T, Candinas D, Beldi G. Biologic mesh implantation is associated with serious abdominal wall complications in patients undergoing emergency abdominal surgery: A randomized-controlled clinical trial. J Trauma Acute Care Surg. 2020 Dec;89(6):1149-1155. doi: 10.1097/TA.0000000000002877. PMID 32649617
- [Derived] Pucciarelli S, Del Bianco P, Pace U, Bianco F, Restivo A, Maretto I, Selvaggi F, Zorcolo L, De Franciscis S, Asteria C, Urso EDL, Cuicchi D, Pellino G, Morpurgo E, La Torre G, Jovine E, Belluco C, La Torre F, Amato A, Chiappa A, Infantino A, Barina A, Spolverato G, Rega D, Kilmartin D, De Salvo GL, Delrio P. Multicentre randomized clinical trial of colonic J pouch or straight stapled colorectal reconstruction after low anterior resection for rectal cancer. Br J Surg. 2019 Aug;106(9):1147-1155. doi: 10.1002/bjs.11222. Epub 2019 Jun 24. PMID 31233220